CLINICAL TRIAL: NCT05375955
Title: A PHASE 2B, RANDOMIZED, DOUBLE BLIND, VEHICLE CONTROLLED, PARALLEL GROUP STUDY TO ASSESS THE EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF MULTIPLE DOSE LEVELS OF PF-07038124 OINTMENT FOR 12 WEEKS IN PARTICIPANTS 12 YEARS AND OLDER AND WITH MILD-TO-MODERATE ATOPIC DERMATITIS OR MILD-TO-SEVERE PLAQUE PSORIASIS
Brief Title: A Study to Learn About The Study Medicine (PF-07038124) In Patients With Mild To Moderate Atopic Dermatitis Or Mild To Severe Plaque Psoriasis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3941005
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis; Plaque Psoriasis
Keywords: Eczema; topical
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Atopic Dermatitis PF-07038124 0.01% ointment (Experimental): Atopic Dermatitis
  Interventions: Drug: PF-07038124 ointment 0.01%
- Atopic Dermatitis Vehicle ointment (Placebo Comparator): Atopic Dermatitis
  Interventions: Drug: Vehicle ointment
- Atopic Dermatitis PF-07038124 0.03% ointment (Experimental): Atopic Dermatitis
  Interventions: Drug: PF-07038124 ointment 0.03%
- Plaque Psoriasis PF-07038124 0.01% ointment (Experimental): Plaque Psoriasis
  Interventions: Drug: PF-07038124 ointment 0.01%
- Plaque Psoriasis PF-07038124 0.03% ointment (Experimental): Plaque Psoriasis
  Interventions: Drug: PF-07038124 ointment 0.03%
- Plaque Psoriasis PF-07038124 0.06% ointment (Experimental): Plaque Psoriasis
  Interventions: Drug: PF-07038124 ointment 0.06%
- Plaque Psoriasis Vehicle ointment (Placebo Comparator): Plaque Psoriasis
  Interventions: Drug: Vehicle ointment

INTERVENTIONS:
Drug: PF-07038124 ointment 0.01% — Atopic Dermatitis and Plaque Psoriasis
  Arms: Atopic Dermatitis PF-07038124 0.01% ointment; Plaque Psoriasis PF-07038124 0.01% ointment
Drug: Vehicle ointment — Atopic Dermatitis and Plaque Psoriasis
  Arms: Atopic Dermatitis Vehicle ointment; Plaque Psoriasis Vehicle ointment
Drug: PF-07038124 ointment 0.03% — Atopic Dermatitis and Plaque Psoriasis
  Arms: Atopic Dermatitis PF-07038124 0.03% ointment; Plaque Psoriasis PF-07038124 0.03% ointment
Drug: PF-07038124 ointment 0.06% — PF-07038124 ointment 0.06% (Plaque Psoriasis only)
  Arms: Plaque Psoriasis PF-07038124 0.06% ointment

SUMMARY:
The purpose of this clinical trial is to learn about the safety, how well the study medicine works, extent to which side effects can be tolerated, and how the study medicine is changed and eliminated from your body after you apply it on your skin. The study medicine is in ointment form.

This study is seeking participants who

If they have Atopic Dermatitis (AD):

* Have a diagnosis for at least 3 months
* Have a diagnosis of mild or moderate disease assessed using Investigator's Global Assessment (IGA)
* Have percent Body Surface Area (%BSA) covering 5% up to 40%
* A Peak Pruritus Numerical Rating Scale (PP-NRS) average score of ≥2 during the screening period

If they have plaque psoriasis (PsO):

* Have a diagnosis for at least 6 months
* Have a diagnosis of mild, moderate, or severe disease assessed using Physician's Global Assessment (PGA)
* Have percent Body Surface Area (%BSA) covering 2% up to 20%

All participants in this study will receive either 0.01% PF-07038124, 0.03% PF-07038124, or a vehicle ointment. In addition, some participants with PsO will receive 0.06% PF- PF-07038124. Participants will not know which dose level they have received. The participants will be randomly assigned to each dose group.

PF-07038124 ointment will be applied topically to affected areas once daily. We will compare the experiences of people receiving the different dose levels of the ointment to those who receive the vehicle ointment. This will help us determine if PF-07038124 ointment is safe and effective.

Participants will take part in this study for approximately 21 weeks. Participants will apply the study medicine once daily for 12 weeks followed by a safety follow-up period of 4-5 weeks from last application of study medicine to last visit.

ELIGIBILITY:
Inclusion Criteria for AD population:

* Diagnosis of Atopic Dermatitis (AD) for at least 3 months
* Investigator's Global Assessment (IGA) score of 2 (mild), or 3 (moderate)
* AD covering 5% and up to 40% of Body Surface Area (BSA)
* A Peak Pruritus Numerical Rating Scale (PP-NRS) average score of ≥2

Inclusion Criteria for Plaque Psoriasis

* Diagnosis of Plaque Psoriasis (PsO) for at least 6 months
* Physician Global Assessment (PGA) score of 2 (mild), 3 (moderate), or 4 (severe)
* PsO covering 2% to 20% (inclusive) of BSA

Exclusion Criteria:

* Presence of skin comorbidities that would interfere with study assessment or response to treatment
* Psychiatric condition including recent or active suicidal ideation or behavior
* Current or recent history of severe, progressive, or uncontrolled disease
* A history of systemic, chronic or acute skin infection requiring hospitalization, parenteral antimicrobial therapy, or is judged clinically significant.
* Recent, significant trauma or major surgery
* History of cancer or have undergone treatment for any type of cancer, with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin or cervical carcinoma in situ with no evidence of recurrence.
* History of angioedema or anaphylaxis to topical products or known sensitivity to any of the components of the investigational products.
* Use of any prohibited concomitant medication(s)
* Previous administration with an investigational drug within 30 days or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* Participants with an estimated glomerular filtration rate (eGFR) of <40 mL/min/1.73m2 calculated using the serum creatinine-based Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) formula for adults and serum creatinine >1.5 x upper limit of normal (ULN) in adolescents (12-18 years old)
* Participants with total bilirubin ≥2x ULN (≥3 x ULN for Gilbert's disease), aspartate aminotransferase (AST) ≥2.5 x ULN, ALT ≥2.5 x ULN.
* Clinically relevant abnormal baseline standard 12-lead electrocardiogram (ECG) including, but not limited to QTC corrected using Fridericia's Formula (QTcF) interval >450 msec and QRS > 120 msec
* A recent history of alcohol or substance abuse

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (22):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Renaissance Research and Medical Group, Cape Coral, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Velocity Clinical Research at The Dermatology Clinic, Baton Rouge, Baton Rouge, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Wayne Health, Dearborn, Michigan
  - Northwell Health Clinical Trials Office, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Health Concepts, Rapid City, South Dakota
  - Clinical Neuroscience Solutions Inc., Memphis, Tennessee
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Memphis, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Canada (7):
  - Dermatology Research Institute, Calgary, Alberta
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research Inc., Markham, Ontario
  - DermEdge Research, Mississauga, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Centre de Recherche Dermatologique du Quebec metropolitain, Québec
- Japan (5):
  - Takagi Dermatological Clinic Branch, Obihiro, Hokkaido
  - Takagi Dermatology, Obihiro, Hokkaido
  - Dermatology Shimizu Clinic, Kobe, Hyōgo
  - Dermatology and Ophthalmology Kume Clinic, Sakai, Osaka
  - Shirasaki dermatology clinic, Takaoka, Toyama
- United Kingdom (3):
  - Egin Research High Wycombe, High Wycombe, Buckinghamshire
  - Southampton General Hospital, Southampton, Hampshire
  - Accellacare - North London, Northwood, London, CITY of

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3941005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 263 participants were enrolled and randomized in the study.
Groups:
- Atopic Dermatitis: Vehicle Ointment: Participants with mild or moderate atopic dermatitis applied the vehicle ointment topically on affected areas once daily (QD) for 12 weeks.
- Atopic Dermatitis: PF-07038124 0.01% Ointment: Participants with mild or moderate atopic dermatitis applied PF-07038124 0.01% ointment topically on affected areas QD for 12 weeks.
- Atopic Dermatitis: PF-07038124 0.03% Ointment: Participants with mild or moderate atopic dermatitis applied PF-07038124 0.03% ointment topically on affected areas QD for 12 weeks.
- Psoriasis: PF-07038124 Vehicle Ointment: Participants with mild, moderate, or severe psoriasis applied PF-07038124 0% ointment topically on affected areas QD for 12 weeks.
- Psoriasis: PF-07038124 0.01% Ointment: Participants with mild, moderate, or severe psoriasis applied PF-07038124 0.01% ointment topically on affected areas QD for 12 weeks.
- Psoriasis: PF-07038124 0.03% Ointment: Participants with mild, moderate, or severe psoriasis applied PF-07038124 0.03% ointment topically on affected areas QD for 12 weeks.
- Psoriasis: PF-07038124 0.06% Ointment: Participants with mild, moderate, or severe psoriasis applied PF-07038124 0.06% ointment topically on affected areas QD for 12 weeks.
Period: Treatment (12 Weeks)
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Started | 44 | 42 | 42 | 34 | 33 | 35 | 33
Treated | 44 | 42 | 42 | 34 | 33 | 35 | 33
Completed | 32 | 34 | 29 | 25 | 28 | 30 | 29
Not Completed | 12 | 8 | 13 | 9 | 5 | 5 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2 | 1 | 1 | 1 | 0
Not completed — Physician Decision | 4 | 1 | 3 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by parent/guardian | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 4 | 7 | 8 | 4 | 3 | 3
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Follow-up (up to 5 Weeks)
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Started | 36 (Participants who discontinued treatment period might enter into follow-up period.) | 36 (Participants who discontinued treatment period might enter into follow-up period.) | 36 (Participants who discontinued treatment period might enter into follow-up period.) | 25 | 28 | 31 (Participants who discontinued treatment period might enter into follow-up period.) | 31 (Participants who discontinued treatment period might enter into follow-up period.)
Completed | 32 | 35 | 31 | 25 | 27 | 29 | 29
Not Completed | 4 | 1 | 5 | 0 | 1 | 2 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician's decision | 2 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention who received at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment | Total
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33 | 263
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (18.55) | 44.1 (15.31) | 40.0 (16.28) | 52.6 (12.28) | 47.8 (13.37) | 55.7 (15.11) | 50.0 (17.33) | 51.6 (14.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 25 | 23 | 14 | 13 | 14 | 15 | 127
  Male | 21 | 17 | 19 | 20 | 20 | 21 | 18 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 11 | 8 | 16 | 11 | 7 | 6 | 66
  Not Hispanic or Latino | 35 | 29 | 32 | 17 | 22 | 25 | 27 | 187
  Unknown or Not Reported | 2 | 2 | 2 | 1 | 0 | 3 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 8 | 8 | 13 | 7 | 4 | 8 | 12 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 13 | 11 | 12 | 0 | 1 | 2 | 0 | 39
  White | 23 | 20 | 17 | 25 | 27 | 25 | 20 | 157
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Investigator's Global Assessment (IGA) Score of Clear (0) or Almost Clear (1) and a Reduction From Baseline of More Than or Equal to (>=) 2 Points at Week 12: Participants With Atopic Dermatitis (AD) Only
Description: IGA assessed severity of AD on 5-point scale ranging from 0(clear)to 4(severe)higher scores indicate more severity,reflecting a global consideration of erythema (ery),induration and scaling. Clinical evaluator assessed overall severity of AD and assigned IGA score as follows: 0 (clear) no inflammatory signs of AD; 1=almost clear, AD not fully cleared-light pink residual lesions(except post-inflammatory hyperpigmentation),just perceptible ery, papulation/induration lichenification, excoriation, no oozing/crusting; 2=mild AD with light red lesions, slight but definite ery, papulation/induration, lichenification, excoriation, no oozing/crusting; 3=moderate AD with red lesions, moderate ery, papulation/induration, lichenification, excoriation, slight oozing/crusting; 4=severe AD with deep dark red lesions, severe ery, papulation/induration, lichenification, excoriation, moderate to severe oozing/crusting.95 percentage (%)confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 12
Population: Intent-to-treat (ITT) analysis set included all participants randomly assigned to study intervention. For this outcome measure (OM), data collection was not planned for the 4 arms of Psoriasis Vehicle QD, Psoriasis PF-07038124 0.01% QD, Psoriasis PF-07038124 0.03% and Psoriasis PF-07038124 0.06% ointment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 44 | 42 | 42
Percentage of participants | 11.4 [4.6 to 24.4] | 23.8 [12.1 to 38.7] | 21.4 [11.4 to 36.4]
Statistical Analysis 1: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Test type: Other; p = 0.0711, Chan and Zhang (1999) method; Risk Difference (RD) = 12.4, 95% CI 2-sided [-4.1 to 29.4]
Statistical Analysis 2: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Test type: Other; p = 0.1290, Chan and Zhang (1999) method; Risk Difference (RD) = 10.1, 95% CI 2-sided [-6.1 to 26.8]

2. Primary Outcome: Percentage of Participants With Physician's Global Assessment (PGA) Score of Clear (0) or Almost Clear (1) and a Reduction From Baseline of >=2 Points at Week 12: Participants With Plaque Psoriasis Only
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). In this OM, percentages of participants with a PGA score of 0 or 1 and an improvement of >=2 from Baseline in PGA score were reported. 95% confidence interval (CI) was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 12
Population: ITT analysis set included all participants randomly assigned to study intervention. For this OM, data collection was not planned for the 3 arms of AD Vehicle QD, AD PF-07038124 0.01% QD and AD PF-07038124 0.03% QD.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 34 | 33 | 35 | 33
Percentage of participants | 8.8 [2.4 to 22.2] | 15.2 [6.2 to 30.8] | 37.1 [21.5 to 55.1] | 45.5 [28.1 to 62.2]
Statistical Analysis 1: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Test type: Other; p = 0.2712, Chan and Zhang (1999) method; Risk Difference (RD) = 6.3, 95% CI 2-sided [-10.8 to 24.3]
Statistical Analysis 2: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Test type: Other; p = 0.0028, Chan and Zhang (1999) method; Risk Difference (RD) = 28.3, 95% CI 2-sided [7.7 to 47.5]
Statistical Analysis 3: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Test type: Other; p = 0.0003, Chan and Zhang (1999) method; Risk Difference (RD) = 36.6, 95% CI 2-sided [14.7 to 56.4]

3. Secondary Outcome: Percentage of Participants With >= 75% Improvement in Eczema Area and Severity Index Total Score (EASI-75) From Baseline, at Week 1, 2, 4, 6, 8, 10, 12: Participants With Atopic Dermatitis Only
Description: EASI quantified severity of AD based on severity of lesion clinical signs and % of body surface area(BSA)affected.Severity of clinical signs of AD lesions (erythema [E], induration/papulation[I],excoriation[Ex] and lichenification[L]) were scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin)], lower limbs [including buttocks]) on a 4-point scale:0= absent; 1= mild;2= moderate;3= severe.EASI area score was based on % BSA with AD in body region: 0(0%), 1(>0 to <10%),2 (10 to <30%), 3(30 to <50%), 4(50 to <70%), 5(70 to <90%) and 6(90 to 100%).Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu)+0.3*At*(Et+It+Ext+Lt)+0.4*Al*(El+Il+Exl+Ll);A= EASI area score;h= head and neck;u= upper limbs;t= trunk;l= lower limbs.Total EASI score=0.0 to 72.0, higher scores indicate greater severity of AD.EASI 75 response was defined as at least a 75% reduction in EASI relative to Baseline.95% CI was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention. For this OM, data collection was not planned for the 4 arms of Psoriasis Vehicle QD, Psoriasis PF-07038124 0.01% QD, Psoriasis PF-07038124 0.03% and Psoriasis PF-07038124 0.06% ointment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 44 | 42 | 42
Percentage of participants
  Week 1 | 2.3 [0.1 to 11.5] | 2.4 [0.1 to 12.1] | 4.8 [0.9 to 15.7]
  Week 2 | 2.3 [0.1 to 11.5] | 11.9 [4.8 to 25.3] | 7.1 [2.0 to 18.7]
  Week 4 | 11.4 [4.6 to 24.4] | 11.9 [4.8 to 25.3] | 16.7 [7.5 to 30.0]
  Week 6 | 13.6 [6.1 to 26.3] | 21.4 [11.4 to 36.4] | 16.7 [7.5 to 30.0]
  Week 8 | 15.9 [7.2 to 29.0] | 19.0 [8.9 to 33.5] | 14.3 [6.4 to 27.7]
  Week 10 | 13.6 [6.1 to 26.3] | 21.4 [11.4 to 36.4] | 19.0 [8.9 to 33.5]
  Week 12 | 13.6 [6.1 to 26.3] | 26.2 [14.9 to 41.0] | 28.6 [15.7 to 43.3]
Statistical Analysis 1: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.5701, Chan and Zhang (1999) method; Risk Difference (RD) = 0.1, 95% CI 2-sided [-10.2 to 10.7]
Statistical Analysis 2: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.3269, Chan and Zhang (1999) method; Risk Difference (RD) = 2.5, 95% CI 2-sided [-8.4 to 14.1]
Statistical Analysis 3: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.0532, Chan and Zhang (1999) method; Risk Difference (RD) = 9.6, 95% CI 2-sided [-2.0 to 23.7]
Statistical Analysis 4: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.1705, Chan and Zhang (1999) method; Risk Difference (RD) = 4.9, 95% CI 2-sided [-6.1 to 17.6]
Statistical Analysis 5: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.5123, Chan and Zhang (1999) method; Risk Difference (RD) = 0.5, 95% CI 2-sided [-14.4 to 15.7]
Statistical Analysis 6: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.3, 95% CI 2-sided [-10.7 to 22.1]
Statistical Analysis 7: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.2736, Chan and Zhang (1999) method; Risk Difference (RD) = 7.8, 95% CI 2-sided [-8.9 to 24.8]
Statistical Analysis 8: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.3967, Chan and Zhang (1999) method; Risk Difference (RD) = 3.0, 95% CI 2-sided [-13.0 to 19.8]
Statistical Analysis 9: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.3997, Chan and Zhang (1999) method; Risk Difference (RD) = 3.1, 95% CI 2-sided [-13.6 to 20.2]
Statistical Analysis 10: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.5461, Chan and Zhang (1999) method; Risk Difference (RD) = -1.6, 95% CI 2-sided [-17.7 to 15.3]
Statistical Analysis 11: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.2736, Chan and Zhang (1999) method; Risk Difference (RD) = 7.8, 95% CI 2-sided [-8.9 to 24.8]
Statistical Analysis 12: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.2754, Chan and Zhang (1999) method; Risk Difference (RD) = 5.4, 95% CI 2-sided [-11.0 to 22.1]
Statistical Analysis 13: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.0977, Chan and Zhang (1999) method; Risk Difference (RD) = 12.6, 95% CI 2-sided [-4.8 to 30.3]
Statistical Analysis 14: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.0542, Chan and Zhang (1999) method; Risk Difference (RD) = 14.9, 95% CI 2-sided [-2.8 to 33.2]

4. Secondary Outcome: Percentage of Participants With >=75% Improvement in Psoriasis Area and Severity Index Total Score (PASI-75) From Baseline, at Week 1, 2, 4, 6, 8, 10, 12: Participants With Plaque Psoriasis Only
Description: The PASI quantified the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI was a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score could vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI score =0.1Ah(Eh+Ih+Sh) + 0.2Au(Eu+Iu+Su) + 0.3At(Et+It+St) + 0.4Al(El+Il+Sl) (A= PASI area score,S=scaling)PASI 75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline. 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 34 | 33 | 35 | 33
Percentage of participants
  Week 1 | 0 [0.0 to 9.0] | 3.0 [0.2 to 15.6] | 0 [0.0 to 8.7] | 9.1 [2.5 to 22.9]
  Week 2 | 0 [0.0 to 9.0] | 9.1 [2.5 to 22.9] | 2.9 [0.1 to 14.6] | 15.2 [6.2 to 30.8]
  Week 4 | 0 [0.0 to 9.0] | 15.2 [6.2 to 30.8] | 14.3 [5.8 to 28.8] | 21.2 [9.2 to 37.8]
  Week 6 | 0 [0.0 to 9.0] | 21.2 [9.2 to 37.8] | 22.9 [11.0 to 39.4] | 33.3 [19.2 to 51.8]
  Week 8 | 2.9 [0.2 to 15.1] | 18.2 [8.2 to 33.8] | 25.7 [13.8 to 42.1] | 33.3 [19.2 to 51.8]
  Week 10 | 8.8 [2.4 to 22.2] | 30.3 [15.6 to 48.2] | 28.6 [14.6 to 44.9] | 48.5 [30.8 to 66.2]
  Week 12 | 14.7 [6.0 to 29.8] | 27.3 [14.7 to 45.1] | 25.7 [13.8 to 42.1] | 51.5 [33.8 to 69.2]
Statistical Analysis 1: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.2578, Chan and Zhang (1999) method; Risk Difference (RD) = 3.0, 95% CI 2-sided [-7.8 to 15.8]
Statistical Analysis 2: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 1.0000, Chan and Zhang (1999) method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-10.6 to 10.1]
Statistical Analysis 3: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 1; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 4: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 5: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.2697, Chan and Zhang (1999) method; Risk Difference (RD) = 2.9, 95% CI 2-sided [-7.8 to 14.9]
Statistical Analysis 6: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 2; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 7: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 8: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.0129, Chan and Zhang (1999) method; Risk Difference (RD) = 14.3, 95% CI 2-sided [2.6 to 30.3]
Statistical Analysis 9: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 4; Test type: Other; p = 0.0024, Chan and Zhang (1999) method; Risk Difference (RD) = 21.2, 95% CI 2-sided [8.0 to 38.9]
Statistical Analysis 10: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.0024, Chan and Zhang (1999) method; Risk Difference (RD) = 21.2, 95% CI 2-sided [8.0 to 38.9]
Statistical Analysis 11: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.0018, Chan and Zhang (1999) method; Risk Difference (RD) = 22.9, 95% CI 2-sided [9.5 to 40.1]
Statistical Analysis 12: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 6; Test type: Other; p = 0.0001, Chan and Zhang (1999) method; Risk Difference (RD) = 33.3, 95% CI 2-sided [17.8 to 51.8]
Statistical Analysis 13: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.0259, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [-0.1 to 32.5]
Statistical Analysis 14: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.0038, Chan and Zhang (1999) method; Risk Difference (RD) = 22.8, 95% CI 2-sided [6.3 to 40.4]
Statistical Analysis 15: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 8; Test type: Other; p = 0.0007, Chan and Zhang (1999) method; Risk Difference (RD) = 30.4, 95% CI 2-sided [12.2 to 48.9]
Statistical Analysis 16: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.0146, Chan and Zhang (1999) method; Risk Difference (RD) = 21.5, 95% CI 2-sided [2.1 to 41.2]
Statistical Analysis 17: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.0205, Chan and Zhang (1999) method; Risk Difference (RD) = 19.7, 95% CI 2-sided [1.0 to 38.9]
Statistical Analysis 18: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 10; Test type: Other; p = 0.0002, Chan and Zhang (1999) method; Risk Difference (RD) = 39.7, 95% CI 2-sided [17.1 to 59.3]
Statistical Analysis 19: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.1245, Chan and Zhang (1999) method; Risk Difference (RD) = 12.6, 95% CI 2-sided [-7.8 to 32.6]
Statistical Analysis 20: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.1431, Chan and Zhang (1999) method; Risk Difference (RD) = 11.0, 95% CI 2-sided [-9.1 to 31.5]
Statistical Analysis 21: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 12; Test type: Other; p = 0.0007, Chan and Zhang (1999) method; Risk Difference (RD) = 36.8, 95% CI 2-sided [12.2 to 56.8]

5. Secondary Outcome: Percentage of Participants With IGA Score of Clear (0) or Almost Clear (1) and a Reduction From Baseline of >= 2 Points at Weeks 1, 2, 4, 6, 8 and 10: Participants With Atopic Dermatitis Only
Description: IGA assessed severity of AD on 5-point scale ranging from 0(clear)to 4(severe)higher scores indicate more severity,reflecting a global consideration of erythema (ery),induration and scaling. Clinical evaluator assessed overall severity of AD and assigned IGA score as follows: 0 (clear) no inflammatory signs of AD; 1=almost clear, AD not fully cleared-light pink residual lesions(except post-inflammatory hyperpigmentation),just perceptible ery, papulation/induration lichenification, excoriation, no oozing/crusting; 2=mild AD with light red lesions, slight but definite ery, papulation/induration, lichenification, excoriation, no oozing/crusting; 3=moderate AD with red lesions, moderate ery, papulation/induration, lichenification, excoriation, slight oozing/crusting; 4=severe AD with deep dark red lesions, severe ery, papulation/induration, lichenification, excoriation, moderate to severe oozing/crusting.95%confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, and 10
Population: ITT analysis set included all participants randomly assigned to study intervention. For this outcome measure (OM), data collection was not planned for the 4 arms of Psoriasis Vehicle QD, Psoriasis PF-07038124 0.01% QD, Psoriasis PF-07038124 0.03% and Psoriasis PF-07038124 0.06% ointment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 44 | 42 | 42
Percentage of participants
  Week 1 | 2.3 [0.1 to 11.5] | 4.8 [0.9 to 15.7] | 4.8 [0.9 to 15.7]
  Week 2 | 2.3 [0.1 to 11.5] | 7.1 [2.0 to 18.7] | 9.5 [3.3 to 21.6]
  Week 4 | 9.1 [3.2 to 20.5] | 14.3 [6.4 to 27.7] | 11.9 [4.8 to 25.3]
  Week 6 | 6.8 [1.9 to 18.6] | 14.3 [6.4 to 27.7] | 14.3 [6.4 to 27.7]
  Week 8 | 6.8 [1.9 to 18.6] | 16.7 [7.5 to 30.0] | 9.5 [3.3 to 21.6]
  Week 10 | 11.4 [4.6 to 24.4] | 19.0 [8.9 to 33.5] | 14.3 [6.4 to 27.7]
Statistical Analysis 1: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.3269, Chan and Zhang (1999) method; Risk Difference (RD) = 2.5, 95% CI 2-sided [-8.4 to 14.1]
Statistical Analysis 2: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.3269, Chan and Zhang (1999) method; Risk Difference (RD) = 2.5, 95% CI 2-sided [-8.4 to 14.1]
Statistical Analysis 3: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.1705, Chan and Zhang (1999) method; Risk Difference (RD) = 4.9, 95% CI 2-sided [-6.1 to 17.6]
Statistical Analysis 4: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.1118, Chan and Zhang (1999) method; Risk Difference (RD) = 7.3, 95% CI 2-sided [-3.9 to 20.5]
Statistical Analysis 5: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.2, 95% CI 2-sided [-9.5 to 20.5]
Statistical Analysis 6: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.3857, Chan and Zhang (1999) method; Risk Difference (RD) = 2.8, 95% CI 2-sided [-11.4 to 17.6]
Statistical Analysis 7: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.1429, Chan and Zhang (1999) method; Risk Difference (RD) = 7.5, 95% CI 2-sided [-6.4 to 22.6]
Statistical Analysis 8: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.1429, Chan and Zhang (1999) method; Risk Difference (RD) = 7.5, 95% CI 2-sided [-6.4 to 22.6]
Statistical Analysis 9: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.1119, Chan and Zhang (1999) method; Risk Difference (RD) = 9.8, 95% CI 2-sided [-4.4 to 25.3]
Statistical Analysis 10: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.3755, Chan and Zhang (1999) method; Risk Difference (RD) = 2.7, 95% CI 2-sided [-10.7 to 16.7]
Statistical Analysis 11: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.2547, Chan and Zhang (1999) method; Risk Difference (RD) = 7.7, 95% CI 2-sided [-8.4 to 24.3]
Statistical Analysis 12: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.3928, Chan and Zhang (1999) method; Risk Difference (RD) = 2.9, 95% CI 2-sided [-12.7 to 18.6]

6. Secondary Outcome: Percentage of Participants With PGA Score of Clear (0) or Almost Clear (1) and a Reduction From Baseline of >=2 Points at Weeks 1, 2, 4, 6, 8 and 10: Participants With Plaque Psoriasis Only
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). In this OM, percentages of participants with a PGA score of 0 or 1 and an improvement of >=2 from Baseline in PGA score were reported. 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, and 10
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 34 | 33 | 35 | 33
Percentage of participants
  Week 1 | 0 [0.0 to 9.0] | 0 [0.0 to 9.2] | 0 [0.0 to 8.7] | 3.0 [0.2 to 15.6]
  Week 2 | 0 [0.0 to 9.0] | 6.1 [1.1 to 19.2] | 5.7 [1.0 to 18.8] | 9.1 [2.5 to 22.9]
  Week 4 | 0 [0.0 to 9.0] | 6.1 [1.1 to 19.2] | 17.1 [7.7 to 32.5] | 15.2 [6.2 to 30.8]
  Week 6 | 0 [0.0 to 9.0] | 15.2 [6.2 to 30.8] | 17.1 [7.7 to 32.5] | 24.2 [11.7 to 42.1]
  Week 8 | 0 [0.0 to 9.0] | 9.1 [2.5 to 22.9] | 28.6 [14.6 to 44.9] | 27.3 [14.7 to 45.1]
  Week 10 | 5.9 [1.1 to 18.8] | 15.2 [6.2 to 30.8] | 31.4 [18.2 to 47.8] | 39.4 [22.9 to 57.9]
Statistical Analysis 1: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 1.0000, Chan and Zhang (1999) method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-10.6 to 11.0]
Statistical Analysis 2: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 1.0000, Chan and Zhang (1999) method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-10.6 to 10.1]
Statistical Analysis 3: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 1; Test type: Other; p = 0.2578, Chan and Zhang (1999) method; Risk Difference (RD) = 3.0, 95% CI 2-sided [-7.8 to 15.8]
Statistical Analysis 4: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.0993, Chan and Zhang (1999) method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-4.9 to 20.7]
Statistical Analysis 5: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.1140, Chan and Zhang (1999) method; Risk Difference (RD) = 5.7, 95% CI 2-sided [-5.3 to 19.2]
Statistical Analysis 6: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 2; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 7: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.0993, Chan and Zhang (1999) method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-4.9 to 20.7]
Statistical Analysis 8: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.0071, Chan and Zhang (1999) method; Risk Difference (RD) = 17.1, 95% CI 2-sided [4.9 to 33.9]
Statistical Analysis 9: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 4; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 10: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 11: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.0071, Chan and Zhang (1999) method; Risk Difference (RD) = 17.1, 95% CI 2-sided [4.9 to 33.9]
Statistical Analysis 12: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 6; Test type: Other; p = 0.0011, Chan and Zhang (1999) method; Risk Difference (RD) = 24.2, 95% CI 2-sided [10.4 to 42.3]
Statistical Analysis 13: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 14: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.0003, Chan and Zhang (1999) method; Risk Difference (RD) = 28.6, 95% CI 2-sided [14.2 to 46.3]
Statistical Analysis 15: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 8; Test type: Other; p = 0.0007, Chan and Zhang (1999) method; Risk Difference (RD) = 27.3, 95% CI 2-sided [12.9 to 45.8]
Statistical Analysis 16: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.1256, Chan and Zhang (1999) method; Risk Difference (RD) = 9.3, 95% CI 2-sided [-6.6 to 26.4]
Statistical Analysis 17: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.0038, Chan and Zhang (1999) method; Risk Difference (RD) = 25.5, 95% CI 2-sided [7.0 to 44.8]
Statistical Analysis 18: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 10; Test type: Other; p = 0.0007, Chan and Zhang (1999) method; Risk Difference (RD) = 33.5, 95% CI 2-sided [12.8 to 52.6]

7. Secondary Outcome: Percentage of Participants With IGA Score of Clear (0) or Almost Clear (1) at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Atopic Dermatitis Only
Description: IGA assessed severity of AD on 5-point scale ranging from 0(clear)to 4(severe)higher scores indicate more severity,reflecting a global consideration of erythema (ery),induration and scaling. Clinical evaluator assessed overall severity of AD and assigned IGA score as follows: 0 (clear) no inflammatory signs of AD; 1=almost clear, AD not fully cleared-light pink residual lesions(except post-inflammatory hyperpigmentation),just perceptible ery, papulation/induration lichenification, excoriation, no oozing/crusting; 2=mild AD with light red lesions, slight but definite ery, papulation/induration, lichenification, excoriation, no oozing/crusting; 3=moderate AD with red lesions, moderate ery, papulation/induration, lichenification, excoriation, slight oozing/crusting; 4=severe AD with deep dark red lesions, severe ery, papulation/induration, lichenification, excoriation, moderate to severe oozing/crusting. 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 44 | 42 | 42
Percentage of participants
  Week 1 | 2.3 [0.1 to 11.5] | 4.8 [0.9 to 15.7] | 4.8 [0.9 to 15.7]
  Week 2 | 4.5 [0.8 to 15.0] | 7.1 [2.0 to 18.7] | 11.9 [4.8 to 25.3]
  Week 4 | 11.4 [4.6 to 24.4] | 16.7 [7.5 to 30.0] | 19.0 [8.9 to 33.5]
  Week 6 | 9.1 [3.2 to 20.5] | 14.3 [6.4 to 27.7] | 21.4 [11.4 to 36.4]
  Week 8 | 11.4 [4.6 to 24.4] | 16.7 [7.5 to 30.0] | 16.7 [7.5 to 30.0]
  Week 10 | 15.9 [7.2 to 29.0] | 19.0 [8.9 to 33.5] | 19.0 [8.9 to 33.5]
  Week 12 | 15.9 [7.2 to 29.0] | 23.8 [12.1 to 38.7] | 28.6 [15.7 to 43.3]
Statistical Analysis 1: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.3269, Chan and Zhang (1999) method; Risk Difference (RD) = 2.5, 95% CI 2-sided [-8.4 to 14.1]
Statistical Analysis 2: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.3269, Chan and Zhang (1999) method; Risk Difference (RD) = 2.5, 95% CI 2-sided [-8.4 to 14.1]
Statistical Analysis 3: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.3585, Chan and Zhang (1999) method; Risk Difference (RD) = 2.6, 95% CI 2-sided [-9.2 to 15.5]
Statistical Analysis 4: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.1290, Chan and Zhang (1999) method; Risk Difference (RD) = 7.4, 95% CI 2-sided [-5.3 to 22.1]
Statistical Analysis 5: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.3, 95% CI 2-sided [-10.7 to 22.1]
Statistical Analysis 6: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.2547, Chan and Zhang (1999) method; Risk Difference (RD) = 7.7, 95% CI 2-sided [-8.4 to 24.3]
Statistical Analysis 7: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.2, 95% CI 2-sided [-9.5 to 20.5]
Statistical Analysis 8: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.0658, Chan and Zhang (1999) method; Risk Difference (RD) = 12.3, 95% CI 2-sided [-3.8 to 28.8]
Statistical Analysis 9: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.3, 95% CI 2-sided [-10.7 to 22.1]
Statistical Analysis 10: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.2751, Chan and Zhang (1999) method; Risk Difference (RD) = 5.3, 95% CI 2-sided [-10.7 to 22.1]
Statistical Analysis 11: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.3997, Chan and Zhang (1999) method; Risk Difference (RD) = 3.1, 95% CI 2-sided [-13.6 to 20.2]
Statistical Analysis 12: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.3997, Chan and Zhang (1999) method; Risk Difference (RD) = 3.1, 95% CI 2-sided [-13.6 to 20.2]
Statistical Analysis 13: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.2736, Chan and Zhang (1999) method; Risk Difference (RD) = 7.9, 95% CI 2-sided [-9.5 to 25.7]
Statistical Analysis 14: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.1119, Chan and Zhang (1999) method; Risk Difference (RD) = 12.7, 95% CI 2-sided [-5.6 to 31.0]

8. Secondary Outcome: Percentage of Participants With PGA Score of Clear (0) or Almost Clear (1) at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Plaque Psoriasis Only
Description: The PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear). 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 34 | 33 | 35 | 33
Percentage of participants
  Week 1 | 0 [0.0 to 9.0] | 0 [0.0 to 9.2] | 2.9 [0.1 to 14.6] | 3.0 [0.2 to 15.6]
  Week 2 | 0 [0.0 to 9.0] | 6.1 [1.1 to 19.2] | 5.7 [1.0 to 18.8] | 9.1 [2.5 to 22.9]
  Week 4 | 0 [0.0 to 9.0] | 6.1 [1.1 to 19.2] | 17.1 [7.7 to 32.5] | 15.2 [6.2 to 30.8]
  Week 6 | 0 [0.0 to 9.0] | 15.2 [6.2 to 30.8] | 17.1 [7.7 to 32.5] | 24.2 [11.7 to 42.1]
  Week 8 | 0 [0.0 to 9.0] | 9.1 [2.5 to 22.9] | 28.6 [14.6 to 44.9] | 27.3 [14.7 to 45.1]
  Week 10 | 8.8 [2.4 to 22.2] | 15.2 [6.2 to 30.8] | 34.3 [19.1 to 52.2] | 39.4 [22.9 to 57.9]
  Week 12 | 11.8 [4.1 to 27.2] | 15.2 [6.2 to 30.8] | 40.0 [25.0 to 57.9] | 45.5 [28.1 to 62.2]
Statistical Analysis 1: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 1.0000, Chan and Zhang (1999) method; Risk Difference (RD) = 0.0, 95% CI 2-sided [-10.6 to 11.0]
Statistical Analysis 2: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.2697, Chan and Zhang (1999) method; Risk Difference (RD) = 2.9, 95% CI 2-sided [-7.8 to 14.9]
Statistical Analysis 3: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 1; Test type: Other; p = 0.2578, Chan and Zhang (1999) method; Risk Difference (RD) = 3.0, 95% CI 2-sided [-7.8 to 15.8]
Statistical Analysis 4: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.0993, Chan and Zhang (1999) method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-4.9 to 20.7]
Statistical Analysis 5: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.1140, Chan and Zhang (1999) method; Risk Difference (RD) = 5.7, 95% CI 2-sided [-5.3 to 19.2]
Statistical Analysis 6: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 2; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 7: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.0993, Chan and Zhang (1999) method; Risk Difference (RD) = 6.1, 95% CI 2-sided [-4.9 to 20.7]
Statistical Analysis 8: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.0071, Chan and Zhang (1999) method; Risk Difference (RD) = 17.1, 95% CI 2-sided [4.9 to 33.9]
Statistical Analysis 9: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 4; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 10: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.0104, Chan and Zhang (1999) method; Risk Difference (RD) = 15.2, 95% CI 2-sided [3.2 to 32.0]
Statistical Analysis 11: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.0071, Chan and Zhang (1999) method; Risk Difference (RD) = 17.1, 95% CI 2-sided [4.9 to 33.9]
Statistical Analysis 12: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 6; Test type: Other; p = 0.0011, Chan and Zhang (1999) method; Risk Difference (RD) = 24.2, 95% CI 2-sided [10.4 to 42.3]
Statistical Analysis 13: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.0436, Chan and Zhang (1999) method; Risk Difference (RD) = 9.1, 95% CI 2-sided [-2.1 to 24.3]
Statistical Analysis 14: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.0003, Chan and Zhang (1999) method; Risk Difference (RD) = 28.6, 95% CI 2-sided [14.2 to 46.3]
Statistical Analysis 15: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 8; Test type: Other; p = 0.0007, Chan and Zhang (1999) method; Risk Difference (RD) = 27.3, 95% CI 2-sided [12.9 to 45.8]
Statistical Analysis 16: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.2712, Chan and Zhang (1999) method; Risk Difference (RD) = 6.3, 95% CI 2-sided [-10.8 to 24.3]
Statistical Analysis 17: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.0056, Chan and Zhang (1999) method; Risk Difference (RD) = 25.5, 95% CI 2-sided [5.4 to 44.8]
Statistical Analysis 18: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 10; Test type: Other; p = 0.0017, Chan and Zhang (1999) method; Risk Difference (RD) = 30.6, 95% CI 2-sided [9.7 to 50.5]
Statistical Analysis 19: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.3929, Chan and Zhang (1999) method; Risk Difference (RD) = 3.4, 95% CI 2-sided [-14.9 to 21.6]
Statistical Analysis 20: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.0040, Chan and Zhang (1999) method; Risk Difference (RD) = 28.2, 95% CI 2-sided [7.0 to 47.7]
Statistical Analysis 21: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 12; Test type: Other; p = 0.0012, Chan and Zhang (1999) method; Risk Difference (RD) = 33.7, 95% CI 2-sided [10.4 to 53.7]

9. Secondary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Atopic Dermatitis Only
Description: EASI quantified severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema [E], induration/papulation [I], excoriation [Ex] and lichenification [L]) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score=0.0 to 72.0, higher scores indicate greater severity of AD. 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention. Here, 'Number Analyzed' signifies participants evaluable for the specified rows. For this OM, data collection was not planned for the 4 arms of Psoriasis Vehicle QD, Psoriasis PF-07038124 0.01% QD, Psoriasis PF-07038124 0.03% and Psoriasis PF-07038124 0.06% ointment.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 44 | 42 | 42
Percent change
  Week 1: number analyzed (Participants) | 40 | 39 | 38
  Week 1 | -10.07 (35.340) | -24.58 (26.168) | -21.07 (27.609)
  Week 2: number analyzed (Participants) | 41 | 40 | 37
  Week 2 | -20.10 (35.277) | -35.91 (28.570) | -35.35 (30.467)
  Week 4: number analyzed (Participants) | 39 | 38 | 38
  Week 4 | -31.06 (37.602) | -47.23 (28.432) | -46.43 (29.199)
  Week 6: number analyzed (Participants) | 35 | 35 | 35
  Week 6 | -33.89 (41.636) | -47.89 (34.117) | -51.96 (32.322)
  Week 8: number analyzed (Participants) | 37 | 37 | 33
  Week 8 | -33.85 (41.950) | -53.67 (30.285) | -53.44 (29.639)
  Week 10: number analyzed (Participants) | 31 | 35 | 31
  Week 10 | -41.88 (39.244) | 55.70 (29.250) | -53.34 (35.171)
  Week 12: number analyzed (Participants) | 34 | 34 | 29
  Week 12 | -36.05 (50.080) | -58.40 (29.835) | -53.29 (38.096)

10. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Total Score at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Plaque Psoriasis Only
Description: The PASI quantified the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI was a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score could vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI =0.1Ah(Eh+Ih+Sh) + 0.2Au(Eu+Iu+Su) + 0.3At(Et+It+St) + 0.4Al(El+Il+Sl) (A= PASI area score,S=scaling)PASI 75 response was defined as at least a 75 percent (%) reduction in PASI relative to Baseline. 95% confidence interval was based on Blyth-Still-Casella method.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable for the specified rows. For this OM, data collection was not planned for the 3 arms of AD Vehicle QD, AD PF-07038124 0.01% QD and AD PF-07038124 0.03% QD.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 34 | 33 | 35 | 33
Units on a scale
  Week 1: number analyzed (Participants) | 29 | 33 | 34 | 30
  Week 1 | -0.60 (1.796) | -1.74 (1.529) | -1.69 (2.053) | -2.66 (2.064)
  Week 2: number analyzed (Participants) | 29 | 32 | 34 | 31
  Week 2 | -1.53 (2.192) | -2.75 (2.315) | -2.41 (2.496) | -3.84 (3.357)
  Week 4: number analyzed (Participants) | 28 | 32 | 33 | 32
  Week 4 | -1.70 (3.245) | -3.09 (2.332) | -3.50 (2.861) | -4.77 (3.694)
  Week 6: number analyzed (Participants) | 23 | 28 | 31 | 29
  Week 6 | -2.13 (3.451) | -3.65 (2.639) | -4.54 (3.143) | -5.39 (3.797)
  Week 8: number analyzed (Participants) | 24 | 29 | 31 | 26
  Week 8 | -3.23 (3.584) | -3.70 (3.059) | -4.73 (3.383) | -6.51 (4.002)
  Week 10: number analyzed (Participants) | 23 | 26 | 31 | 29
  Week 10 | -3.93 (3.398) | -4.45 (3.486) | -4.87 (3.369) | -5.74 (3.973)
  Week 12: number analyzed (Participants) | 25 | 28 | 31 | 29
  Week 12 | -3.57 (3.946) | -4.53 (3.556) | -4.84 (3.530) | -6.07 (4.058)

11. Secondary Outcome: Percentage of Participants With >= 4 Points of Reduction From Baseline in Weekly Average of Peak Pruritus Numerical Rating Scale (PP-NRS) at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Atopic Dermatitis Only
Description: The PP-NRS was a daily participant reported assessment of intensity of pruritus on an 11-point numerical rating scale ranging from 0 ('No Itch) to 10 ('Worst Itch Imaginable'), with a 24-hour recall period. Participants were asked to assess their itch intensity over the past 24 hours, on a scale from 0 (no itching) to 10 (worst possible itching). Higher scores indicated worse itch. For the PP-NRS score, baseline was defined as the average of all values recorded between Day -7 (7 days prior to dosing) and Day -1 (1 day prior to dosing). In this OM, percentages of AD participants with >=4 points of reduction in weekly averages of PP-NRS from baseline are reported (percentage based on number of participants with baseline >=4).
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. For this outcome measure (OM), data collection was not planned for the 4 arms of Psoriasis Vehicle QD, Psoriasis PF-07038124 0.01% QD, Psoriasis PF-07038124 0.03% and Psoriasis PF-07038124 0.06% ointment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment
Number analyzed (Participants) | 40 | 38 | 34
Percentage of participants
  Week 1 | 2.5 [0.1 to 12.7] | 5.3 [0.9 to 17.5] | 0 [0.0 to 9.0]
  Week 2 | 0 [0.0 to 7.8] | 18.4 [8.1 to 33.4] | 14.7 [6.0 to 29.8]
  Week 4 | 10.0 [3.5 to 22.7] | 23.7 [12.7 to 38.9] | 29.4 [15.1 to 46.5]
  Week 6 | 17.5 [7.8 to 31.5] | 21.1 [10.0 to 35.8] | 26.5 [14.3 to 43.6]
  Week 8 | 17.5 [7.8 to 31.5] | 21.1 [10.0 to 35.8] | 29.4 [15.1 to 46.5]
  Week 10 | 17.5 [7.8 to 31.5] | 23.7 [12.7 to 38.9] | 26.5 [14.3 to 43.6]
  Week 12 | 15.0 [6.7 to 29.3] | 26.3 [13.4 to 42.1] | 35.3 [20.0 to 53.5]
Statistical Analysis 1: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.3255, Chan and Zhang (1999) method; Risk Difference (RD) = 2.8, 95% CI 2-sided [-8.5 to 15.8]
Statistical Analysis 2: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.7181, Chan and Zhang (1999) method; Risk Difference (RD) = -2.5, 95% CI 2-sided [-13.3 to 8.3]
Statistical Analysis 3: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.0022, Chan and Zhang (1999) method; Risk Difference (RD) = 18.4, 95% CI 2-sided [7.0 to 34.3]
Statistical Analysis 4: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.0064, Chan and Zhang (1999) method; Risk Difference (RD) = 14.7, 95% CI 2-sided [3.7 to 31.1]
Statistical Analysis 5: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.0659, Chan and Zhang (1999) method; Risk Difference (RD) = 13.7, 95% CI 2-sided [-3.4 to 31.5]
Statistical Analysis 6: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.0189, Chan and Zhang (1999) method; Risk Difference (RD) = 19.4, 95% CI 2-sided [0.9 to 38.5]
Statistical Analysis 7: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.3962, Chan and Zhang (1999) method; Risk Difference (RD) = 3.6, 95% CI 2-sided [-14.9 to 22.3]
Statistical Analysis 8: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.2333, Chan and Zhang (1999) method; Risk Difference (RD) = 9.0, 95% CI 2-sided [-10.4 to 29.1]
Statistical Analysis 9: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.3962, Chan and Zhang (1999) method; Risk Difference (RD) = 3.6, 95% CI 2-sided [-14.9 to 22.3]
Statistical Analysis 10: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.1353, Chan and Zhang (1999) method; Risk Difference (RD) = 11.9, 95% CI 2-sided [-7.9 to 32.7]
Statistical Analysis 11: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.2791, Chan and Zhang (1999) method; Risk Difference (RD) = 6.2, 95% CI 2-sided [-12.8 to 25.7]
Statistical Analysis 12: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.2333, Chan and Zhang (1999) method; Risk Difference (RD) = 9.0, 95% CI 2-sided [-10.4 to 29.1]
Statistical Analysis 13: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.1295, Chan and Zhang (1999) method; Risk Difference (RD) = 11.3, 95% CI 2-sided [-7.3 to 30.6]
Statistical Analysis 14: Comparison: Atopic Dermatitis: Vehicle Ointment vs Atopic Dermatitis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.0247, Chan and Zhang (1999) method; Risk Difference (RD) = 20.3, 95% CI 2-sided [0.1 to 40.2]

12. Secondary Outcome: Percentage of Adult (18-75 Years Old) Participants With >=4 Points of Reduction From Baseline in Weekly Average of PP-NRS at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Plaque Psoriasis Only
Description: The PP-NRS was a daily participant reported assessment of intensity of pruritus on an 11-point numerical rating scale ranging from 0 ('No Itch) to 10 ('Worst Itch Imaginable'), with a 24-hour recall period. Participants were asked to assess their itch intensity over the past 24 hours, on a scale from 0 (no itching) to 10 (worst possible itching). Higher scores indicated worse itch. For the PP-NRS score, baseline was defined as the average of all values recorded between Day -7 (7 days prior to dosing) and Day -1 (1 day prior to dosing). In this OM, percentages of plaque psoriasis participants (18-75 years old) with >=4 points of reduction in weekly averages of PP-NRS from baseline are reported (percentage based on number of participants with baseline >=4).
Time Frame: Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention.Here,'Overall Number of Participants Analyzed'=participants evaluable for this OM,all participants reported under'Overall Number of Participants Analyzed'contributed data to table but may not have evaluable data for every row.Here,'Number Analyzed'=participants evaluable for specified rows.For this OM,data collection was not planned for 3 arms:AD Vehicle QD, PF-07038124 0.01% QD,AD PF-07038124 0.03% QD ointment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 33 | 33 | 31 | 31
Percentage of participants
  Week 1: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 1 | 4.3 [0.2 to 19.8] | 0 [0.0 to 13.9] | 12.5 [3.5 to 30.8] | 5.3 [0.3 to 24.4]
  Week 2: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 2 | 4.3 [0.2 to 19.8] | 13.6 [3.8 to 32.6] | 20.8 [8.6 to 40.6] | 21.1 [7.5 to 43.4]
  Week 4: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 4 | 8.7 [1.6 to 26.8] | 22.7 [9.4 to 45.1] | 25.0 [11.5 to 44.7] | 26.3 [11.0 to 50.0]
  Week 6: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 6 | 4.3 [0.2 to 19.8] | 31.8 [13.9 to 54.9] | 25.0 [11.5 to 44.7] | 42.1 [22.2 to 65.5]
  Week 8: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 8 | 17.4 [6.2 to 38.5] | 40.9 [20.7 to 61.7] | 25.0 [11.5 to 44.7] | 52.6 [31.2 to 75.6]
  Week 10: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 10 | 17.4 [6.2 to 38.5] | 36.4 [18.7 to 58.2] | 29.2 [12.6 to 50.0] | 47.4 [24.4 to 68.8]
  Week 12: number analyzed (Participants) | 23 | 22 | 24 | 19
  Week 12 | 17.4 [6.2 to 38.5] | 40.9 [20.7 to 61.7] | 33.3 [16.9 to 55.3] | 47.4 [24.4 to 68.8]
Statistical Analysis 1: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 1; Test type: Other; p = 0.7278, Chan and Zhang (1999) method; Risk Difference (RD) = -4.3, 95% CI 2-sided [-21.9 to 11.5]
Statistical Analysis 2: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 1; Test type: Other; p = 0.2548, Chan and Zhang (1999) method; Risk Difference (RD) = 8.2, 95% CI 2-sided [-11.5 to 28.2]
Statistical Analysis 3: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 1; Test type: Other; p = 0.5162, Chan and Zhang (1999) method; Risk Difference (RD) = 0.9, 95% CI 2-sided [-17.5 to 21.9]
Statistical Analysis 4: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 2; Test type: Other; p = 0.1663, Chan and Zhang (1999) method; Risk Difference (RD) = 9.3, 95% CI 2-sided [-11.4 to 30.7]
Statistical Analysis 5: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 2; Test type: Other; p = 0.0605, Chan and Zhang (1999) method; Risk Difference (RD) = 16.5, 95% CI 2-sided [-4.2 to 38.3]
Statistical Analysis 6: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 2; Test type: Other; p = 0.0592, Chan and Zhang (1999) method; Risk Difference (RD) = 16.7, 95% CI 2-sided [-5.4 to 41.6]
Statistical Analysis 7: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 4; Test type: Other; p = 0.1246, Chan and Zhang (1999) method; Risk Difference (RD) = 14.0, 95% CI 2-sided [-8.6 to 37.4]
Statistical Analysis 8: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 4; Test type: Other; p = 0.0789, Chan and Zhang (1999) method; Risk Difference (RD) = 16.3, 95% CI 2-sided [-7.3 to 39.7]
Statistical Analysis 9: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 4; Test type: Other; p = 0.0889, Chan and Zhang (1999) method; Risk Difference (RD) = 17.6, 95% CI 2-sided [-6.4 to 43.7]
Statistical Analysis 10: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 6; Test type: Other; p = 0.0097, Chan and Zhang (1999) method; Risk Difference (RD) = 27.5, 95% CI 2-sided [4.2 to 50.7]
Statistical Analysis 11: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 6; Test type: Other; p = 0.0294, Chan and Zhang (1999) method; Risk Difference (RD) = 20.7, 95% CI 2-sided [-0.8 to 43.6]
Statistical Analysis 12: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 6; Test type: Other; p = 0.0018, Chan and Zhang (1999) method; Risk Difference (RD) = 37.8, 95% CI 2-sided [10.9 to 62.2]
Statistical Analysis 13: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 8; Test type: Other; p = 0.0495, Chan and Zhang (1999) method; Risk Difference (RD) = 23.5, 95% CI 2-sided [-3.8 to 48.9]
Statistical Analysis 14: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 8; Test type: Other; p = 0.2890, Chan and Zhang (1999) method; Risk Difference (RD) = 7.6, 95% CI 2-sided [-17.3 to 32.4]
Statistical Analysis 15: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 8; Test type: Other; p = 0.0103, Chan and Zhang (1999) method; Risk Difference (RD) = 35.2, 95% CI 2-sided [5.1 to 62.0]
Statistical Analysis 16: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 10; Test type: Other; p = 0.1088, Chan and Zhang (1999) method; Risk Difference (RD) = 19.0, 95% CI 2-sided [-7.8 to 44.8]
Statistical Analysis 17: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 10; Test type: Other; p = 0.2719, Chan and Zhang (1999) method; Risk Difference (RD) = 11.8, 95% CI 2-sided [-14.0 to 36.2]
Statistical Analysis 18: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 10; Test type: Other; p = 0.0227, Chan and Zhang (1999) method; Risk Difference (RD) = 30.0, 95% CI 2-sided [0.4 to 56.6]
Statistical Analysis 19: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.01% Ointment; Week 12; Test type: Other; p = 0.0495, Chan and Zhang (1999) method; Risk Difference (RD) = 23.5, 95% CI 2-sided [-3.8 to 48.9]
Statistical Analysis 20: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.03% Ointment; Week 12; Test type: Other; p = 0.1246, Chan and Zhang (1999) method; Risk Difference (RD) = 15.9, 95% CI 2-sided [-10.6 to 40.6]
Statistical Analysis 21: Comparison: Psoriasis: PF-07038124 Vehicle Ointment vs Psoriasis: PF-07038124 0.06% Ointment; Week 12; Test type: Other; p = 0.0227, Chan and Zhang (1999) method; Risk Difference (RD) = 30.0, 95% CI 2-sided [0.4 to 56.6]

13. Secondary Outcome: Percent Change From Baseline in Affected Body Surface Area (BSA) at Weeks 1, 2, 4, 6, 8, 10 and 12: Participants With Atopic Dermatitis and Plaque Psoriasis
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall percentage (%) BSA for individuals with AD ranged from 5-40 % BSA and for individuals with Psoriasis ranged from 2-20 % BSA. Higher % BSA = greater area affected.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: ITT analysis set included all participants randomly assigned to study intervention. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable for the specified timepoints.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Percent change
  Week 1: number analyzed (Participants) | 40 | 39 | 38 | 29 | 33 | 34 | 30
  Week 1 | -5.70 (21.189) | -7.97 (20.319) | -11.34 (27.214) | -0.57 (3.095) | -11.80 (22.429) | -4.08 (24.592) | -11.24 (23.946)
  Week 2: number analyzed (Participants) | 41 | 40 | 37 | 29 | 32 | 34 | 31
  Week 2 | -7.71 (38.699) | -19.19 (26.809) | -25.17 (33.618) | -0.09 (19.604) | -20.88 (30.731) | -9.60 (31.828) | -20.62 (26.613)
  Week 4: number analyzed (Participants) | 39 | 38 | 38 | 28 | 32 | 33 | 32
  Week 4 | -23.51 (42.066) | -30.05 (32.224) | -36.52 (36.063) | 3.14 (27.814) | -24.40 (33.837) | -23.27 (33.581) | -33.16 (32.929)
  Week 6: number analyzed (Participants) | 35 | 35 | 35 | 23 | 28 | 31 | 29
  Week 6 | -20.81 (38.584) | -33.20 (37.302) | -41.40 (39.631) | 1.19 (23.562) | -36.37 (37.798) | -30.76 (33.598) | -44.91 (38.196)
  Week 8: number analyzed (Participants) | 37 | 37 | 33 | 24 | 29 | 31 | 26
  Week 8 | -21.12 (49.459) | -35.81 (34.333) | -43.59 (39.783) | 0.75 (30.196) | -31.98 (47.562) | -34.04 (38.481) | -51.30 (39.210)
  Week 10: number analyzed (Participants) | 31 | 35 | 31 | 23 | 26 | 31 | 29
  Week 10 | -27.68 (44.681) | -36.84 (36.966) | -36.38 (50.533) | -3.77 (26.271) | -42.72 (47.305) | 36.35 (38.176) | -49.14 (38.319)
  Week 12: number analyzed (Participants) | 34 | 34 | 29 | 25 | 28 | 31 | 29
  Week 12 | -19.45 (48.697) | -40.87 (41.005) | -46.53 (44.420) | -7.61 (42.825) | -38.16 (48.923) | -36.13 (39.779) | -60.83 (39.223)

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs): Participants With Atopic Dermatitis and Plaque Psoriasis
Description: An AE was any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered TEAE if the event occurred on or after the first dosing date but before the last dose plus the lag time (35 days).
Time Frame: From start of study treatment up to 35 days after last dose of treatment (up to 19 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants | 20 | 28 | 19 | 9 | 13 | 11 | 19

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs): Participants With Atopic Dermatitis and Plaque Psoriasis
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; resulted in congenital anomaly/birth defect, was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or other important medical events.
Time Frame: From start of study treatment up to 35 days after last dose of treatment (up to 19 weeks)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants | 0 | 1 | 1 | 0 | 0 | 0 | 1

16. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs: Participants With Atopic Dermatitis and Plaque Psoriasis
Description: Temperature, pulse rate, and blood pressure were assessed in vital sign examination. Body temperature was collected using oral, tympanic, axillary or temporal methods. Blood pressure and pulse rate measurements were assessed with the participant in a supine or seated position using a completely automated device after at least 5 minutes of rest for the participant. Clinically significant changes were determined by the investigator.
Time Frame: From start of study treatment (Day 1) up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG): Participants With Atopic Dermatitis and Plaque Psoriasis
Description: A standard 12-lead ECG utilizing limb leads was collected using ECG machine that automatically calculated the heart rate and measured pulse rate, QT, and QTc intervals and QRS complex. Clinically significant findings (including, but not limited to, changes from baseline in QTcF after enrollment) were determined by the investigator or qualified designee.
Time Frame: From start of study treatment (Day 1) up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants With Laboratory Abnormalities: Participants With Atopic Dermatitis and Plaque Psoriasis
Description: Laboratory assessments included hematology, clinical chemistry and urinalysis. Clinically significant abnormal laboratory findings were those which were not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: From start of study treatment (Day 1) up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants | 18 | 27 | 18 | 14 | 14 | 13 | 15

19. Secondary Outcome: Number of Participants According to Worst Severity Grades in Local Skin Tolerability: Participants With Atopic Dermatitis and Plaque Psoriasis
Description: The investigator or designee assessed tolerability at the site of study intervention application, immediately post-application of the study intervention. Skin Tolerability Grading System for non-lesional skin included grade 0 (No evidence of local intolerance), grade 1 (Mild-Minimal erythema and/or edema, slight glazed appearance), grade 2 (Moderate-Definite erythema and/or edema with peeling and/or cracking but needs no adaptation of posology), grade 3 (Severe-Erythema, edema glazing with fissures, few vesicles or papules: consider removing topical agent [if still in place], grade 4 (very severe- Strong reaction spreading beyond the treated area, bullous reaction, erosions: removal of topical agent [if still in place].
Time Frame: From start of study treatment (Day 1) up to Week 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
Number analyzed (Participants) | 44 | 42 | 42 | 34 | 33 | 35 | 33
Participants
  Grade 0 (None) | 44 | 42 | 42 | 32 | 32 | 34 | 33
  Grade 1 (Mild) | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Grade 2 (Moderate) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 (Severe) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4 (Very severe) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 35 days after last dose of treatment (up to 19 weeks)
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in 1 participant and as non-serious in another participant, or 1 participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Atopic Dermatitis: Vehicle Ointment | Atopic Dermatitis: PF-07038124 0.01% Ointment | Atopic Dermatitis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 Vehicle Ointment | Psoriasis: PF-07038124 0.01% Ointment | Psoriasis: PF-07038124 0.03% Ointment | Psoriasis: PF-07038124 0.06% Ointment
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/42 | 0/42 | 0/34 | 0/33 | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/44 | 1/42 | 1/42 | 0/34 | 0/33 | 0/35 | 1/33
Other Adverse Events (participants affected / at risk) | 0/44 | 5/42 | 2/42 | 1/34 | 5/33 | 2/35 | 7/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atopic Dermatitis: Vehicle Ointment (N=44) | Atopic Dermatitis: PF-07038124 0.01% Ointment (N=42) | Atopic Dermatitis: PF-07038124 0.03% Ointment (N=42) | Psoriasis: PF-07038124 Vehicle Ointment (N=34) | Psoriasis: PF-07038124 0.01% Ointment (N=33) | Psoriasis: PF-07038124 0.03% Ointment (N=35) | Psoriasis: PF-07038124 0.06% Ointment (N=33)
Pancreatic mass (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atopic Dermatitis: Vehicle Ointment (N=44) | Atopic Dermatitis: PF-07038124 0.01% Ointment (N=42) | Atopic Dermatitis: PF-07038124 0.03% Ointment (N=42) | Psoriasis: PF-07038124 Vehicle Ointment (N=34) | Psoriasis: PF-07038124 0.01% Ointment (N=33) | Psoriasis: PF-07038124 0.03% Ointment (N=35) | Psoriasis: PF-07038124 0.06% Ointment (N=33)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 5 | 2 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT05375955/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT05375955/SAP_001.pdf